CLINICAL TRIAL: NCT02964078
Title: Coordinated High Dose Interleukin-2 (Aldesleukin, Proleukin™) and Pembrolizumab (Anti-PD1, Keytruda™) for Therapy of Metastatic Kidney Cancer
Brief Title: Interleukin-2 and Pembrolizumab for Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Prometheus Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18536; MISP# 52587 (Other: Merck); IIT15PLK02 (Other: Prometheus Laboratories)
Record Dates: First submitted 2016-11-11; First posted 2016-11-15 (Estimated); Results first posted 2020-04-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Kidney Cancer
Keywords: Kidney Disease; Metastatic; Antibody
MeSH Terms: conditions — Kidney Neoplasms; Kidney Diseases; Neoplasm Metastasis | interventions — pembrolizumab; spartalizumab; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and Interleukin-2 (Experimental): Outpatient Intravenous (IV) infusion of Pembrolizumab and Inpatient IV infusion of Interleukin-2.
  Interventions: Drug: Pembrolizumab; Drug: Interleukin-2

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab: 200 mg every 3 weeks, 12 doses planned. This is considered the investigational part of the combination. The infusion time is 1 hour.
  Other Names: anti-PD-1 antibody; Keytruda™
Drug: Interleukin-2 — Interleukin-2: 8 admissions to hospital, each with 5 doses planned. This is considered the standard part of the combination. The standard interleukin-2 dose is 600,000 international units per kilogram per dose, with a maximum of 66,000,000 (for patients over 110 kg, which is 242 pounds). The dose is usually set at the start of the treatment and not adjusted. The infusion time is 15 minutes.
  Other Names: aldesleukin; Proleukin™; IL-2

SUMMARY:
The main purpose of this study is to evaluate the effects of the interleukin-2 given in combination with pembrolizumab.

Interleukin-2 (IL-2) is also called aldesleukin, or Proleukin™.

Pembrolizumab is also called Keytruda™, or anti-PD-1 antibody.

DETAILED DESCRIPTION:
The treatment is organized into blocks of 9 weeks, with pembrolizumab treatment planned for weeks 1, 4 and 7. On the second and third blocks, interleukin-2 is added, for 5 doses at a time, one dose every 8 hours, on a weekly schedule on the two weeks after the week 1 and the week 4 pembrolizumab doses.

There is no dose escalation portion: The dose and schedule of IL-2 is fixed, 600,000 IU/kg/dose, with a cap of 66 mIU/dose. Doses may be omitted for safety. The dose of pembrolizumab is fixed, flat dose 200 mg/dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis/Condition for Entry into the Trial: Metastatic kidney cancer. Clear cell histology component from primary or metastatic lesion.
* Willing and able to provide written informed consent for the trial.
* Age over 18 on day of signing informed consent.
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Willing to provide tissue from a newly obtained or archival tissue, if available.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function, as outlined in Table 1 of study protocol document.
* Females of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Females of childbearing potential must agree to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
* Males must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Cardiac testing with either exercise stress test or thallium stress test, within 3 months of start of the first treatment day. Atrial fibrillation that is rate controlled is allowed. Note - the first treatment day is about 9 weeks before the first IL-2 treatment day. If a cardiologist's evaluation determines that this is superfluous based on other assessments, then this may be omitted.
* Pulmonary function test is required, within 3 months of start.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active Bacillus Tuberculosis (TB).
* Has hypersensitivity to pembrolizumab or any of its excipients.
* The number of prior therapies is restricted as follows: (a) Zero or one prior therapies during the preceding one year. This serves to limit the treatment cohort to patients with either only slowly progressive disease, or up to one prior therapy. (b) No prior PD-1 or PD-L1 antibody therapies are allowed. (c) Prior IL-2 is allowed, if it finished more than 1 year prior. (d) The following are not counted as medical therapies: nephrectomy, radiation therapy, other energy-ablative techniques, or metastasectomy.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. - Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. - Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Potential participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment that would be exclusionary.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., hepatitis C virus (HCV) RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Myocardial infarction, stroke, coronary artery bypass surgery, coronary stent, or unstable angina within one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2025-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Chatzkel, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab and Interleukin-2
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab and Interleukin-2
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall Response According to Immune-related response criteria (irRC). Overall response rate ORR is defined with confirmation of the response status Complete Response (CR) or Partial Response (PR) among the combination treatment population patients; the binomial estimate and its one-sided 95% confidence interval will be reported. CR: Disappearance of all lesions in two consecutive observation not less than 4 weeks apart. PR: ≥50% decrease in tumor burden compared with baseline in two observations at least 4 weeks apart.
Time Frame: Up to 24 months
Measure: Median (90% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab and Interleukin-2
Number analyzed (Participants) | 27
percentage of participants | 70.4 [54.6 to 100]

2. Secondary Outcome: Overall Survival (OS) of Intent to Treat (ITT) Population
Description: Analysis: Overall Survival (OS) of ITT patients using Kaplan-Meier estimate, counting from the eligible date to death from any cause, or censored on end of known follow up, either within this study or in the Prometheus Laboratories sponsored PROCLAIM registry (PROCLAIM Registry to Evaluate the Treatment Patterns and Clinical Response in Malignancy, NCT01415167).
Time Frame: Up to 24 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pembrolizumab and Interleukin-2
Number analyzed (Participants) | 27
proportion of participants | 1 [.871 to 1]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) of ITT patients using Kaplan Meier estimate, from the confirmed eligible date to the first occurrence of disease progression or death, from any cause, or lost to follow up, whichever is earliest; or censored at last follow-up during study. Progressive Disease (PD): At least 25% increase in tumor burden compared with nadir (at any single time point) in two consecutive observations at least 4 weeks apart.
Time Frame: Up to 24 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pembrolizumab and Interleukin-2
Number analyzed (Participants) | 27
proportion of participants | .630 [.421 to .781]

ADVERSE EVENTS:
Time Frame: Adverse events recorded from Cycle 1 day 1 through 30 days after cessation of treatment
Arm/Group | Pembrolizumab and Interleukin-2
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 17/27
Other Adverse Events (participants affected / at risk) | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and Interleukin-2 (N=27)
Atrial fibrilation (Cardiac disorders) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Flu like symptoms (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Creatinine increased (Investigations) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 4 (8)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Edema cerebral (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 2 (4)
Acute kidney injury (Renal and urinary disorders) | 6 (6)
Renal and urinary disorders - Other (Renal and urinary disorders) | 8 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 7 (12)
Blood bilirubin increased (Investigations) | 3 (4)
Renal and urinary disorders - Other (Renal and urinary disorders) | 8 (8)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Lymphocyte count decreased (Investigations) | 7 (19)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (14)
Hypertension (Vascular disorders) | 3 (6)
Vascular disorders - Other (Vascular disorders) | 2 (3)
Leukocytosis (Blood and lymphatic system disorders) | 5 (10)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and Interleukin-2 (N=27)
Creatinine increased (Investigations) | 7 (12)
Lymphocyte count decreased (Investigations) | 7 (19)
Blood bilirubin increased (Investigations) | 5 (6)
Urine output decreased (Investigations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2)
Investigations - Other (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (14)
Hyponatremia (Metabolism and nutrition disorders) | 5 (9)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hyperalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 8 (10)
Atrial fibrillation (Cardiac disorders) | 4 (5)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Asystole (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (6)
Hypertension (Vascular disorders) | 4 (8)
Capillary leak syndrome (Vascular disorders) | 3 (3)
Vascular disorders - Other (Vascular disorders) | 2 (2)
Renal and urinary disorders - Other (Renal and urinary disorders) | 6 (7)
Acute kidney injury (Renal and urinary disorders) | 6 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Skin and subcutaneous tissue disorders -Other (Skin and subcutaneous tissue disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 3 (4)
Edema limbs (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
General disorders and administration site conditions -Other (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 6 (10)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (5)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Infections and Infestations - Other (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT02964078/Prot_SAP_000.pdf